CLINICAL TRIAL: NCT06191978
Title: A Phase Ia/Ib Open-label, Multiple Dose, Study to Determine the Recommended Dose, Evaluate PKs, PDs, Safety, and Activity of Venetoclax in Combination With Oral Decitabine/Cedazuridine (ASTX727) in Pediatric Patients With Relapsed/Refractory Acute Myeloid Leukemia (AML)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0661; NCI-2023-10826 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — decitabine and cedazuridine drug combination; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ASTX727/venetoclax (Experimental): On Days 1-5 of Cycle 1, you will take ASTX727 by mouth with a glass of water. Participants must fast (not eat or drink anything but water, black coffee, or tea) for at least 2 hours before and for 2 hours after taking ASTX727. For 4 hours before dosing and 4 hours after dosing, participants should not take antacids or any other medicine that can change the amount of acid in your stomach.
  Days 1-21 or 1-28 depending on dose level, of all cycles beginning with Cycle 2. The study doctor will tell participants which of these schedules participants will follow. Venetoclax should be taken with water and a meal at around the same time each day.
  Interventions: Drug: ASTX727; Drug: Venetoclax

INTERVENTIONS:
Drug: ASTX727 — Given by PO
  Other Names: Inqovi
Drug: Venetoclax — Given by PO
  Other Names: ABT-199; GDC-0199

SUMMARY:
To find a recommended dose of ASTX727 (cedazuridine/decitabine) in combination with venetoclax for pediatric patients with relapsed AML.

DETAILED DESCRIPTION:
Primary Objectives

1. To determine the recommended dose of ASTX727 when given in combination with venetoclax in relapsed/refractory (R/R) pediatric participants with acute myeloid leukemia (AML).
2. To evaluate and describe the toxicities of ASTX727 and venetoclax administered in R/R AML pediatric population.
3. To characterize the pharmacokinetic (PK) and pharmacodynamic (PD) profile of ASTX727 alone and in combination with venetoclax in an R/R AML pediatric population.

Secondary Objectives

1. To evaluate the potential for drug-drug interactions: effect of venetoclax on PK of ASTX727.
2. To define preliminary efficacy of ASTX727 when given in combination with venetoclax in pediatric participants. Efficacy will be based on Best Overall Response (BOR), including complete remission (CR), CR with incomplete blood count recovery, CR with incomplete hematologic recovery), and partial remission, overall survival (OS), event-free survival (EFS), and duration of response (DOR) of pediatric participants treated with this combination.

Exploratory Objectives To quantify the number of pediatric participants transitioning to Hematopoietic stem cell transplant (HSCT), i.e., CR/CRi/CRh rate, HR.

To identify biological markers of response to venetoclax and/or its combination with ASTX727. These effects could be at the molecular, cellular, or cytogenetic level.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric Participants with Relapsed/refractory AML by WHO criteria.
2. Participants must have ≥ 5% blasts in the bone marrow as assessed by morphology or flow cytometry. However, if an adequate bone marrow sample cannot be obtained, participants may be enrolled if there is unequivocal evidence of leukemia with ≥ 5% blasts in the peripheral blood or an AML defining genetic abnormality as specified by the WHO 2022 criteria.
3. Performance status: Lansky ≥ 50 for participants who are ≤ 16 years old and Karnofsky ≥ 50% for participants who are > 16 years old.
4. Age ≥2 years of age and ≤18 years of age
5. Able to swallow pills
6. The following baseline laboratory data:

   1. Total serum bilirubin ≤1.5 x upper limit of normal (ULN) for age. Participants with known Gilbert's syndrome may have a total bilirubin up to ≤5 x ULN for age.
   2. Creatinine clearance (Schwartz-Formula) or radioisotope GFR ≥ 60ml/min/1.73 m2 or a serum creatinine based on age/sex as follows:
   3. Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≤3 x ULN; ≤5 x ULN in case of suspected leukemic liver involvement.
   4. Females of childbearing potential must have a negative serum or urine beta human chorionic gonadotropin (β-HCG) pregnancy test result within 14 days prior to the first dose of study drugs and must agree to use one of the following effective contraception methods during the study and for 6 months following the last dose of study drug. Effective methods of birth control include:

   i. Birth control pills, skin patches, shots, implants (placed under the skin by a health care provider) ii. Intrauterine devices (IUDs) iii. Condom or occlusive cap (diaphragm or cervical/vault caps) used with Spermicide iv. Abstinence e. Males, need to inform the doctor right away if the partner becomes pregnant or suspects pregnancy. While in this study and for 3 months after the last treatment the patient should not donate sperm for the purposes of reproduction. He will need to use a condom while in this study and for 3 months after the last treatment.
7. At least one parents or LAR must provide signature of informed consent and there must be documentation of assent by the subject, as age appropriate, before completing any study-related procedures.

Exclusion Criteria:

1. Concomitant other anti-cancer therapy and/or participation in any other investigational clinical trials except for hydroxyurea. Concurrent hydroxyurea use should be limited to the first 2 cycles of therapy only.
2. History of another primary invasive malignancy that has not been definitively treated and is in remission. Participants with non-melanoma skin cancers or with carcinomas in situ are eligible regardless of the time from diagnosis (including concomitant diagnoses).
3. Presence of clinically significant uncontrolled central nervous system (CNS) pathology such as epilepsy, childhood seizure, paresis, aphasia, stroke, severe brain injuries, organic brain syndrome, or psychosis.
4. Evidence of active cerebral/meningeal disease. Participants may have history of CNS leukemic involvement if definitively treated with prior therapy and no evidence of active disease at the time of consent with at least 2 consecutive spinal fluid negative assessments for residual leukemia and negative imaging (imaging required only if previously showing evidence of CNS leukemia not otherwise documented by spinal fluid assessment).
5. Participants with uncontrolled, active infections (viral, bacterial, or fungal) or other disease expected to interfere with the ability of the PI to assess the efficacy of the study drug. Infections controlled on concurrent anti-microbial agents are acceptable, and anti-microbial prophylaxis per institutional guidelines are acceptable.
6. Known active hepatitis B (eg, HBsAg reactive), or hepatitis C (eg, HCV RNA [qualitative] is detected), or chronic hepatitis B or C infection or human immunodeficiency virus (HIV) infection in medical history, with the following exceptions:

   a. Those with a history of hepatitis with a negative polymerase chain reaction (either qualitative or quantitative) OR have documentation of stable disease with aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase and alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase <2.0×upper limit of normal (ULN) may be eligible for this study.

   b) Subjects with history of HIV who have an undetectable viral load for the prior 3 months, and who agree to maintain antiviral therapy, may be eligible for the study.
7. Liver cirrhosis or other serious active liver disease or with suspected active alcohol abuse.
8. Exclude participants with active GVHD and those on immunosuppressive drugs for treatment of GVHD. Require that participants be off calcineurin inhibitors for at least 4 weeks to be eligible.
9. Prior chemotherapy/radiotherapy/investigational therapy within 2 weeks before the start of study drugs with the following exception:

   a. To reduce the circulating blast count or palliation: intravenous cytarabine, steroids or hydroxyurea. No washout necessary for these agents.
10. Females who are pregnant or lactating.
11. Male or female subjects of childbearing potential, unwilling to use an approved, effective means of contraception.
12. Other severe, uncontrolled acute or chronic medical or psychiatric condition or laboratory abnormality that in the opinion of the Investigator may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and/or would make the participant inappropriate for enrollment into this study.
13. Participants with acute promyelocytic leukemia, juvenile myelomonocytic leukemia, or bone marrow failure syndromes are not eligible.
14. Known or suspected hypersensitivity to decitabine, cedazuridine, or venetoclax.
15. Participants on concomitant medications known to be metabolized by CDA will need review of the medication and assessment of possible impact of avoiding dosing during the 24 hours prior to possible enrollment, at the time of cedazuridine exposure, and 24 hours following the last dose of oral decitabine/cedazuridine.
16. Participants of adult age (= 18 years of age) who are cognitively impaired will not be eligible for this study.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | Through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Amber Gibson, DO, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org